CLINICAL TRIAL: NCT05330936
Title: Comparison of Cyanocobalamin in Avocado Oil Cream With Steroid Combination Ointment in the Treatment of Chronic Plaque Psoriasi-A Randomized Clinical Trial in Tertiary Care Hospital
Brief Title: Comparison of Cyanocobalamin in Avocado Oil Cream With Steroid Combination Ointment
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Pak Emirates Military Hospital (Other)
Responsible Party: Principal Investigator, Ishtiaq Ahmed, Registrar Dermatology, Pak Emirates Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PakEmiratesMH
Record Dates: First submitted 2022-03-23; First posted 2022-04-15 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): Steroid combination ointment in the treatment of chronic Plaque Psoriasis
  Interventions: Combination Product: Potent topical steroid
- Group B (Active Comparator): Cyanocobalamin in Avocado Oil cream in the treatment of chronic Plaque
  Interventions: Combination Product: Potent topical steroid

INTERVENTIONS:
Combination Product: Potent topical steroid — Cyanocobalamin in Avocado Oil Cream

SUMMARY:
A randomized clinical trial with two groups. Group A Group B Group A is being treated with conventional Steroid combination ointment for the treatment of chronic Plaque Psoriasis.

Group B is being treated with Cyanocobalamin in Avocado Oil cream for the treatment of chronic Plaque Psoriasis.

Each group having 45 patients.

DETAILED DESCRIPTION:
Outcome is being measured by PASI Score calculation with monthly follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age bracket (18-60 years)
* Non psoriatic Arthritis
* No oral Retinoids

Exclusion Criteria:

* pregnancy
* Malignancy
* Body surface area involving >50%

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Efficacy and tolerability of steroids as compared to Avacado Oil Cream | 12 weeks
  Compariaon of Efficacy of Steroid combination ointment in the treatment of chronic Plaque Psoriasis

CONTACTS AND LOCATIONS:
Overall Officials: Qamar ud din Khan, MBBS,FCPS, Study Director — Pak Emirates Military Hospital
Locations (1):
- PakEmiratesMH, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No